CLINICAL TRIAL: NCT06998875
Title: A Prospective Cohort Study on the Efficacy and Safety Comparison of Tofacitinib Citrate Tablets Combined With Acitretin Capsules Versus Acitretin Capsules Alone in the Treatment of Primary Cutaneous Amyloidosis
Brief Title: A Prospective Cohort Study on Primary Cutaneous Amyloidosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Army Medical University, China (Other)
Responsible Party: Principal Investigator, Rui Yin, Professor/Chief Physician, Army Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2025060
Record Dates: First submitted 2025-04-13; First posted 2025-05-31 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Primary Cutaneous Amyloidosis
MeSH Terms: conditions — Amyloidosis, Primary Cutaneous | interventions — tofacitinib; Acitretin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Take oral Acitretin capsules, 10mg each time, twice a day, for a continuous period of 16 weeks; at the same time, take Tofactinib tablets, 5mg each time, twice a day, for a continuous period of 16 weeks.
  Interventions: Drug: Tofacitinib and Acitretin Capsules.
- Control group (Active Comparator): Take oral Acitretin capsules, 10mg each time, twice a day, for a continuous course of 16 weeks.
  Interventions: Drug: Acitretin Capsules.

INTERVENTIONS:
Drug: Tofacitinib and Acitretin Capsules. — The same with Arms.
  Arms: Experimental group
Drug: Acitretin Capsules. — The same with Arms.
  Arms: Control group

SUMMARY:
The aim of this clinical trial is to find out whether the combination of tocilizumab tablets and acitretin capsules is more effective than acitretin capsules alone in treating primary cutaneous amyloidosis. It will also investigate the safety of the combination of tocilizumab tablets and acitretin capsules. The main questions it aims to answer are:

1. Does the combination of tocilizumab tablets and acitretin capsules relieve the pruritus symptoms of the participants faster and reduce the pruritus score more than acitretin capsules alone?
2. What medical problems will the participants encounter when taking tocilizumab tablets combined with acitretin capsules? The researchers compared the combination of tocilizumab tablets and acitretin capsules with acitretin capsules alone to see if the combination could better treat primary cutaneous amyloidosis without causing serious adverse reactions.

Participants will:

1. Take the combination of tocilizumab tablets and acitretin capsules or acitretin capsules alone every day for 16 weeks.
2. Visit the clinic once every 4 weeks for checkups and tests.
3. Observe participants at 4 weeks, 12 weeks and 24 weeks after discontinuation of medication to determine the recurrence status.
4. Collect the visual analogue scale (VAS) scores for pruritus, symptom severity (SCORAD) scores , rash area and severity, treatment response (EASI) scores, dermatological quality of life index (DLQI), and insomnia severity index (ISI) of participants before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, without infectious diseases such as "hepatitis B" and "tuberculosis" and major underlying diseases (gender not limited);

  * "Outpatient Diagnosis" includes "primary cutaneous amyloidosis", "macular amyloidosis" or "lichen amyloidosis";

    * Visited the outpatient department for PCA treatment for 4 times or more;

      * The medication record shows "Avastin Capsules" and/or "Tofacitinib Citrate";

        * The medical record fully records baseline characteristics, medication dosage, efficacy assessment and adverse events.

Exclusion Criteria:

* Nodular amyloidosis or combined with other types of amyloidosis (such as systemic amyloidosis);

  * During the study period, other immunosuppressants (such as glucocorticoids, methotrexate) or biologics were used;

    * Incomplete medical records such as demographic data, laboratory parameters, prescription administration and patient prognosis, as well as irregular treatment, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) scores for pruritus. | Week 0, Week 4, Week 8, Week 12 and Week 16.
  The average percentage changes in the visual analogue scale (VAS) scores for pruritus from baseline to Week 4, 8, 12 and 16 after medication administration. VAS score for pruritus ranges from 0 to 10, and the higher the score, the worse the outcome.

SECONDARY OUTCOMES:
SCORAD index. | Week 0, Week 4, Week 8, Week 12 and Week 16.
  SCORAD (Scoring Atopic Dermatitis) Index ranges from 0 to 83, which is used to describe symptoms and signs, and the higher the csore, the more severe the disease.
EASI Index. | Week 0, Week 4, Week 8, Week 12 and Week 16.
  EASI (Eczema area and severity) Index ranges from 0 to 72, which is used to describe the area and severity of the rash and the treatment response, and the higher the score, the larger the area and severity of the rash, and the worse the treatment response.
DLQI. | Week 0, Week 4, Week 8, Week 12 and Week 16.
  DLQI (Dermatology Life Quality Index) ranges from 0 to 30, and the higher the score, the greater the impact on daily life.
ISI. | Week 0, Week 4, Week 8, Week 12 and Week 16.
  ISI (Insomnia Severity Index) ranges from 0 to 28, and the higher the score, the more severe the degree of insomnia.
The onset time of drug efficacy. | Up to 8 weeks.
  When the participants return for follow-up visit, the time elapsed from the moment the participants first started taking the medicine to the point when the symptoms have alleviated or disappeared is calculated.
Recurrence rate. | Within 24 weeks after the treatment concludes.
  Within 24 weeks after the treatment concludes, check whether the participants have any recurrence of the disease.
Incidence rate of adverse events. | Week 4, Week 8, Week 16 and Week 20.
  Liver or kidney function impairment; Abnormal lipid metabolism; Abnormal thyroid function, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Yin, MD, Principal Investigator — Department of Dermatology, Southwest Hospital, Third Military Medical University (Army Medical University)
Locations (1):
- Department of Dermatology, Southwest Hospital, Third Military Medical University (Army Medical University), Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No